CLINICAL TRIAL: NCT05645848
Title: The Rate and Predictors of Vaginal Bleeding Among Women With Placenta Previa: A Cross-sectional Study
Brief Title: The Rate and Predictors of Vaginal Bleeding Among Women With Placenta Previa
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ismail Omar Mohammed Ali, principal investigator, Assiut University
Other Study IDs: placenta previa bleeding rate
Record Dates: First submitted 2022-11-04; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Placenta Previa; Vaginal Bleeding; Antepartum Hemorrhage
MeSH Terms: conditions — Placenta Previa; Uterine Hemorrhage | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasonography — Abdominal ultrasound in pregnant women with placenta previa

SUMMARY:
Placenta previa is usually diagnosed when the placenta implanted in the lower uterine segment, thus partially or totally overlying the internal os . It occurs with an incidence of 0.3-0.5%. It is associated mainly with prior caesarean delivery . The condition is frequently complicated by invasion of placental villi beyond the decidua basalis causing placenta accreta . Placenta previa is a major cause of massive haemorrhage during pregnancy and after delivery . The antepartum bleeding from placenta previa- can be life-threatening, thus, the prediction of this bleeding is of great importance . It is important to distinguish between women at high and low risk for antepartum haemorrhage with placenta previa especially at late pregnancy . However, the potential risk factors for antepartum haemorrhage in women with placenta previa have not been thoroughly examined.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 28 weeks.
* Diagnosed to have placenta previa by ultrasound

Exclusion Criteria:

* Women with complicated pregnancies (e.g. preeclampsia, diabetes mellitus and cardiac, renal, antiphospholipid syndrome).
* Women with premature rupture of membrane.
* Women who will refuse to participate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: pregnant women with placenta previa
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The rate of vaginal bleeding in women presented by placenta previa at third trimester of pregnancy. | Through study completion, an average of 1 and half year
  The rate of vaginal bleeding in women presented by placenta previa at third trimester of pregnancy.

SECONDARY OUTCOMES:
Identification of the potential clinical and ultrasonographic predictors of antepartum hemorrhage in women with placenta previa at third trimester of pregnancy | through study completion, an average of 1 and half year
  The result that the investigators will get from the study will help identify predictors of antepartum hemorrhage in pregnant women with placenta previa and hence preventing it, antepartum hemorrhage is a major life threatening complication of the disease wether to the baby or the mother

CONTACTS AND LOCATIONS:
Overall Officials: Kamal M Zahran, professor, Study Chair — department of obstetrics and gynecology, faculty of medicine, Assuit University, Egypt; Mohamed K Ali, doctor, Study Director — department of obstetrics and gynecology, faculty of medicine, Assuit University, Egypt; Mohamed M Abd-allah, doctor, Study Director — department of obstetrics and gynecology, faculty of medicine, Assuit University, Egypt; Ismael O Ali, resident, Principal Investigator — department of obstetrics and gynecology, faculty of medicine, Assuit University, Egypt

REFERENCES:
- [Background] Wu S, Kocherginsky M, Hibbard JU. Abnormal placentation: twenty-year analysis. Am J Obstet Gynecol. 2005 May;192(5):1458-61. doi: 10.1016/j.ajog.2004.12.074. PMID 15902137
- [Background] Shaamash AH, Ali MK, Attyia KM. Intramuscular 17alpha-hydroxyprogesterone caproate to decrease preterm delivery in women with placenta praevia: a randomised controlled trial. J Obstet Gynaecol. 2020 Jul;40(5):633-638. doi: 10.1080/01443615.2019.1645099. Epub 2019 Oct 31. PMID 31670998
- [Background] Shazly SA, Badee AY, Ali MK. The use of multiple 8 compression suturing as a novel procedure to preserve fertility in patients with placenta accreta: case series. Aust N Z J Obstet Gynaecol. 2012 Aug;52(4):395-9. doi: 10.1111/j.1479-828X.2012.01449.x. Epub 2012 Jun 9. PMID 22681562
- [Background] Nagase Y, Matsuzaki S, Endo M, Hara T, Okada A, Mimura K, Hiramatsu K, Kakigano A, Nakatsuka E, Miyake T, Takiuchi T, Ueda Y, Tomimatsu T, Kimura T. Placenta previa with posterior extrauterine adhesion: clinical features and management practice. BMC Surg. 2021 Jan 6;21(1):10. doi: 10.1186/s12893-020-01027-9. PMID 33407322
- [Background] Dashe JS. Toward consistent terminology of placental location. Semin Perinatol. 2013 Oct;37(5):375-9. doi: 10.1053/j.semperi.2013.06.017. PMID 24176163
- [Background] Love CD, Fernando KJ, Sargent L, Hughes RG. Major placenta praevia should not preclude out-patient management. Eur J Obstet Gynecol Reprod Biol. 2004 Nov 10;117(1):24-9. doi: 10.1016/j.ejogrb.2003.10.039. PMID 15474239